CLINICAL TRIAL: NCT04515446
Title: Sequential Quantification of Viral Load in the Upper Respiratory Tract in Adult Patients Admitted for Influenza and Treated With Olsetamivir
Brief Title: Quantification of Viral Load in the Upper Respiratory Tract in Patients Treated With Olsetamivir for Influenza
Acronym: VIRIDAE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-06
Record Dates: First submitted 2020-01-07; First posted 2020-08-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Flu
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, transversal, diagnostic measurement, blind, descriptive study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TROD + PCR diagnosis (Other): For each patient positive for flu with a rapid diagnostic test, sequential nasopharyngeal (NP) samples will be collected for quantitative PCR every day from D1 to D8 or until discharge (if before D8). Sequential quantitative PCR will quantify influenza virus load in the upper airways.
  Interventions: Diagnostic Test: Rapid test for diagnosis orientation; Diagnostic Test: quantitative PCR

INTERVENTIONS:
Diagnostic Test: Rapid test for diagnosis orientation — Rapid tests screen for influenza viruses in less than 30 minutes. They detect internal viral nucleoproteins by immunochromatography using specific antibodies attached to one or more strips.
  Other Names: TROD
Diagnostic Test: quantitative PCR — Molecular biology method of gene amplification in vitro. It allows a large number of known DNA or RNA sequences to be duplicated

SUMMARY:
Seasonal influenza is a frequent disorder with high impact on morbidity and mortality and significant burden on healthcare-related cost. In France, the 2018-2019 flu epidemic has led to 13,100 all-cause death including 9,900 death directly related to the viral infection.

As cross-transmission of influenza is responsible for nosocomial outbreaks, preventing transmission of infectious agents in healthcare settings is a major issue. If vaccination of patients and healthcare givers remains cornerstone, control procedures are mandatory. Therefore patients admitted with influenza require isolation precautions including admission in a single room and protective measures. Based on experts advise, isolation is currently recommended for 5 to 8 days. Duration of isolation depends on immune status and antiviral therapy. However, during periods of epidemic, every hospital room is valuable and each ressource has to be tightly used. Risk of contamination is related to the presence of influenza in the upper airways. To the Promoteur 's knowledge, presence of influenza in the upper airways has not been studied in patients receiving oseltamivir. The question is : Do duration of isolation in patients admitted with flu decreas when they are treated with antiviral therapy. To answer this question The Promoteur would aim to determine influenza carriage in the upper airways in in-patients treated by olsetamivir.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Positive testing for influenza (A or B)
* Patients hospitalized and treated with olsetamivir
* Signature of informed consent
* Affiliation to healthcare insurance (France, Monaco)

Exclusion Criteria:

* Refusal to participate
* Admission to intensive care
* Palliative care
* Unable to give inform consent
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
The duration of influenza virus carriage in the upper airways in patients treated with olsetamivir will be observed | Within 8 days following patient's participation

SECONDARY OUTCOMES:
Duration of influenza virus carriage in the upper airways among patients treated with olsetamivir according to the viral strand (A or B) will be mesured | Within 8 days following patient's participation
Duration of influenza virus carriage in the upper airways among patients treated with olsetamivir according to their vaccination status and comorbidities will be mesured and compared | Within 8 days following patient's participation
Difference in the number of days in isolation in patients hospitalized and treated with olsetamivir will be evaluated | 21 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Municipality of Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No
no data sharing is planned

REFERENCES:
- [Result] Li X, Zhang Z, Yu A, Ho SY, Carr MJ, Zheng W, Zhang Y, Zhu C, Lei F, Shi W. Global and local persistence of influenza A(H5N1) virus. Emerg Infect Dis. 2014 Aug;20(8):1287-95. doi: 10.3201/eid2008.130910. PMID 25061965
- [Result] Keeler SP, Dalton MS, Cressler AM, Berghaus RD, Stallknecht DE. Abiotic factors affecting the persistence of avian influenza virus in surface waters of waterfowl habitats. Appl Environ Microbiol. 2014 May;80(9):2910-7. doi: 10.1128/AEM.03790-13. Epub 2014 Feb 28. PMID 24584247
- [Result] Patterson Ross Z, Komadina N, Deng YM, Spirason N, Kelly HA, Sullivan SG, Barr IG, Holmes EC. Inter-Seasonal Influenza is Characterized by Extended Virus Transmission and Persistence. PLoS Pathog. 2015 Jun 24;11(6):e1004991. doi: 10.1371/journal.ppat.1004991. eCollection 2015 Jun. PMID 26107631